CLINICAL TRIAL: NCT01526460
Title: Prospective, Randomized, Single Center, Open Label Study Designed to Evaluate the Effect on Platelet Reactivity in Response to High Doses of Atorvastatin or Rosuvastatin Administered Before Percutaneous Coronary Intervention (PCI)
Brief Title: Evaluation of Platelet Function After Statin Loading Dose in Patients Before Percutaneous Coronary Intervention
Acronym: STATIPLAT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Antonio Colombo, MD, IRCCS San Raffaele
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STATIPLAT
Record Dates: First submitted 2011-09-14; First posted 2012-02-03 (Estimated); Last update posted 2014-03-06 (Estimated); Status verified 2014-03

CONDITIONS: Platelet Dysfunction
Keywords: Platelet; Atorvastatin; Rosuvastatin; Multiplate; reactivity
MeSH Terms: interventions — Atorvastatin; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Atorvastatin (Active Comparator): Atorvastatin 80 mg
  Interventions: Drug: Atorvastatin
- Rosuvastatin (Active Comparator): Rosuvastatin 40 mg
  Interventions: Drug: Rosuvastatin
- No statin loading dose (Placebo Comparator): No statin loading dose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Atorvastatin — 80 mg
  Other Names: TORVAST; TOTALIP
  Arms: Atorvastatin
Drug: Rosuvastatin — 40 mg
  Other Names: CRESTOR
  Arms: Rosuvastatin
Drug: Placebo — no statin loading dose
  Other Names: NO STATIN DRUGS
  Arms: No statin loading dose

SUMMARY:
The purpose of this study is to evaluate the effect of a loading dose of two different statins on platelet reactivity (atorvastatin, metabolized by CYP3A4, and rosuvastatin, which is rather independent of this enzyme)in patients at least 5 days in therapy with aspirin and clopidogrel (with or without an undergoing treatment with statins) undergoing PCI for coronary disease with chronic stable angina and/or evidence of inducible myocardial ischemia.

DETAILED DESCRIPTION:
An initial assessment of platelet reactivity in response to the TRAP (thrombin receptor agonist), ADP and arachidonic acid (respectively, indicative of the response to clopidogrel and aspirin) will be performed with impedance aggregometry (Multiplate® analyzer system). Patients with a increased residual platelet reactivity to ADP test (AUC > 47) will receive a different antiplatelet therapy and will then be excluded from the study, the other will be randomized to 3 groups of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-75 years
* Patients with chronic stable angina
* Patients with coronary artery disease or with de novo stent restenosis of native vessels.
* Patients who are able to understand the significance of this study and to adhere to recruitment by signing the informed consent.

Exclusion Criteria:

* Acute Coronary Syndromes with an enzymatic movement (STEMI, NSTEMI).
* Allergy or intolerance to atorvastatin, rosuvastatin, aspirin, clopidogrel.
* Altered basal level of transaminase or CPK.
* Patient with history of hepatitis-acute/chronic.
* Patients already receiving high-dose statins.
* Contraindications to antiplatelet therapy.
* Patients with acute inflammatory disease and/or underlying chronic (hepatitis, pneumonia, urinary tract, rectum ulcerative colitis etc.).
* Patients with anemia (haemoglobin <8.5 mg/dl), leukocytosis (WBC> 12.000 mm3), leukopenia (WBC <3000 mm3), platelet count <100.000; hypersplenism.
* Patients with malignant disease.
* Patients enrolled in other studies not yet completed.
* Patients with known allergy / intolerance to statins.
* Pregnant women and women who are breastfeeding.
* Patients with myopathy (muscle pain and unexplained repeated)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2011-08; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Area Under the Aggregation Curve (AUC) measured with the Multiplate 5.0 Analyzer | Evaluation of platelet reactivity (in terms of AUC) two time points.
  Evaluation of the effect of a loading dose (LD) of two different statins on platelet reactivity (atorvastatin and rosuvastatin) in terms of difference between AUC value before statin LD and after 12 hrs statin LD. The Area Under the Aggregation Curve (AUC) will be measured with the Multiplate 5.0 system.

SECONDARY OUTCOMES:
Incidence of periprocedural myocardial infarction | CK and CK-MB evaluated before the procedure and two time points up to 12 hours
  To evaluate if the loading dose of statin prevent the periprocedural myocardial damage measured by CK and CK-MB The measurments will be done once before the procedure and at 6 and 12 hours after.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Colombo, MD, Principal Investigator — IRCCS San Raffaele Monte Tabor
Locations (1):
- IRCCS San Raffaele Monte Tabor, Milan, Italy